CLINICAL TRIAL: NCT06333132
Title: Deciphering the Role of Incretin Hormones in Weight Loss-induced Remission of Type 2 Diabetes
Brief Title: Deciphering the Role of Incretin Hormones in Weight Loss-induced Remission of Type 2 Diabetes (DIABeat)
Acronym: DiabEATit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Andrea Natali, Professor, Azienda Ospedaliero, Universitaria Pisana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DiabEAT.it
Record Dates: First submitted 2024-03-13; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Diabetes Mellitus Type 2 in Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese subjects with type 2 diabetes mellitus (Experimental): Individualized weight-loss nutritional intervention
  Interventions: Behavioral: Weight loss-induced Diabetes Remission

INTERVENTIONS:
Behavioral: Weight loss-induced Diabetes Remission — Patients will undergo a dietary intervention plus drugs (if needed) with the purpose to obtain a 10% (or at least 10 kg) body weight reduction to achieve diabetes remission

SUMMARY:
The goal of this mechanistic study is to investigate the role of incretin hormones on weight loss-induced type 2 diabetes remission.

DETAILED DESCRIPTION:
Participants will undergo an intensive, individualized dietary treatment to achieve a 10% reduction in body weight, during which glucose-lowering therapy will be withdrawn. Before and after the intervention, the patients will undergo:

* measurement of fasting glucose and glycated hemoglobin
* Indirect calorimetry
* oral glucose tolerance test
* intravenous glucose tolerance test
* quality of life and diet-related questionnaires
* 72-hour food records

At the end of the protocol, subjects will be followed up to maintain lifestyle changes and intercept cases of diabetes relapse.

ELIGIBILITY:
Inclusion Criteria:

* T2D for less than 6 years;
* age 18-65 years;
* both genders;
* BMI 27-45 kg/m2;
* HbA1c 48-108 mmol/mol (43-108 mmol/mol if on glucose-lowering drugs).

Exclusion Criteria:

* type 1 or secondary/genetic diabetes;
* treatment with insulin, Glucagon-Like Peptide-1 agonists, Gastric Inhibitory Peptide/GLP-1 co-agonists, or pioglitazone;
* weight loss >5% within the previous 6 months;
* eGFR <30 ml/min/1.73m2;
* myocardial infarction within the previous 6 months;
* severe heart failure (NYHA III-IV); eating disorder; substance abuse;
* severe depression;
* known cancer;
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with incretin effect's restoration after achieving weightloss-induced diabetes remission | 12 weeks
  The investigators will test whether diabetes remission obtained after 10% weight-loss, induced by an intensive nutritional intervention, is associated with an improvement of the incretin effect from baseline.
  Diabetes remission will be defined according to the latest international consensus as an HbA1c <48 mmol/mol measured at least 3 months after cessation of glucose-lowering pharmacotherapy.
  The restoration of the incretin effect will be assessed by measuring both incretin levels and estimated incretin mediated insulin secretion before and after achieving the weight loss during an Oral Glucose Tolerance Test followed by an intravenous Glucose Tolerance Test.

SECONDARY OUTCOMES:
Rate of sustained weightloss-induced diabetes remission assessed by 2 consecutive HbA1c <48mmol/mol within 6 months | 36 weeks
  Diabetes remission will be defined according to the latest international consensus as an HbA1c <48 mmol/mol measured at least 3 months after cessation of glucose-lowering pharmacotherapy.
  Thus, diabetes remission will be assessed after the end of the intervention phase (V1). Participants who will achieve diabetes remission at V1 will be monitored by measuring HbA1c for the next 6 months at 3-month intervals (V2 and V3).

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Tricò, MD, PhD, Principal Investigator — University of Pisa
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No